CLINICAL TRIAL: NCT05166083
Title: Investigation of the Perceptual and Acoustic Characteristic of Voice in Trans Man
Brief Title: Investigation of the Perceptual and Acoustic Voice in Trans Man
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERVE OGULMUS UYSAL, Principal Investigator, Hacettepe University
Other Study IDs: HUSLPTRANSMANVOICE
Record Dates: First submitted 2021-11-13; First posted 2021-12-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-03

CONDITIONS: Gender Dysphoria; Voice Disorder Due to Transsexualism; Transgender Persons; Hormone Replacement Therapy
Keywords: Trans man voice, hormon therapy
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trans man: "Trans man" is assigned female at birth and identify as man
  Interventions: Other: Testosterone Hormon Therapy

INTERVENTIONS:
Other: Testosterone Hormon Therapy — Testosterone isocaproate, ... ml, 8 doses, once per 21 days

SUMMARY:
The aim of the study is to follow acoustic and perceptual voice changes in trans men during hormone therapy and to examine the relationship between psychosocial and vocal characteristics and testosterone measured in routine follow-up in accordance with international follow-up guidelines.

DETAILED DESCRIPTION:
Trans men who have completed the evaluation and follow-up procedure and decided to use sex hormones will be included in the study. Participants will be followed for 8 doses of sex hormone use. Acoustic and perceptual changes in voice will be monitored at baseline (before hormone use), 4th dose, and 8th dose. The relationship between testosterone and psychosocial and vocal characteristics will be examined. At the baseline of the study, participants will be evaluated with Videolaryngostroboscopy (VLS). As a result of VLS, perceptual and acoustic voice evaluation will be made to the participants who are determined to have healthy vocal folds. During routine psychiatric visits, participants will be asked to fill in self-report scales. Endocrinological routine evaluations will be applied to the participants and the data of these routine evaluations will be used in the study. All of these evaluations (perceptual and acoustic voice evaluation, endocrinological and psychiatric evaluations) will be repeated at the 4. and 8. doses of the hormone therapy, except for the VLS evaluation.

IBM SPSS Statistics 26.0 and Microsoft Excel 365 programs will be used for statistical analysis. The number of participants to be included in the study was calculated using the G Power 3.1 program. In the analysis, the number of participants was determined as 28 (G power=0.80, α =0.05). The normal distribution of the data will be examined by visual and analytical methods (Shapiro-Wilk test, Kolmogorov-Smirnov test).The analysis of each variable measured at three time points will be evaluated using ANOVA if the assumptions of parametric tests are met, and using the Friedman test if the assumptions of parametric tests are not met. When the parametric conditions are met Paired t test will be used to compare the measurement values, and when the parametric conditions are not met, the Wilcoxon signed-rank test will be used. Multiple Regression Analysis will be used to determine the factors affecting the person's own perception of voince. Finally, statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with "Gender Dysphoria" according to DSM 5
* Having decided to start hormone therapy

Exclusion Criteria:

* Diagnosis of vocal fold lesion in videolaryngostroboscopy evaluation
* Having previously received voice therapy or undergone voice surgery
* Having a systematic/or neurological disorder that may affect voice quality
* Having had hormone therapy or still on hormone therapy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — "Trans man" is a person whose assigned sex at birth is female and who identifies himself as male.
Study Population: Trans men who are followed in Hacettepe University Hospital Endocrinology and Psychiatry Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Self-perception of voice | change from baseline to the 4th dose of hormone treatment
  Transsexual Voice Questionnaire (TVQ-Female to male) Score Self-perception of voice masculinity (SPVM) Score
Change in Self-perception of voice | change from baseline to the 8th dose of hormone treatment
  Transsexual Voice Questionnaire (TVQ-Female to male) Score Self-perception of voice masculinity (SPVM) Score
Change in Self-perception of voice | change from 4th to the 8th dose of hormone treatment
  Transsexual Voice Questionnaire (TVQ-Female to male) Score Self-perception of voice masculinity (SPVM) Score

SECONDARY OUTCOMES:
Change in Acoustic Voice Characteristics | change from baseline to the 4th dose of hormone treatment
  Digital recordings will be made using the Computerized Speech Lab (KayPENTAX) while performing the following tasks: sustained vowel /a:/, sponteous speech and "Pinokyo passage" reading. Voice recordings will be analyzed using the Real-Time Pitch Program and the Multidimensional Voice Program for measure F0, Mean F0, Jitter percent, Shimmer Percent, and noise-to-harmonic ratio (NHR).
Change in Acoustic Voice Characteristics | change from baseline to the 8th dose of hormone treatment
  Digital recordings will be made using the Computerized Speech Lab (KayPENTAX) while performing the following tasks: sustained vowel /a:/, sponteous speech and "Pinokyo passage" reading. Voice recordings will be analyzed using the Real-Time Pitch Program and the Multidimensional Voice Program for measure F0, Mean F0, Jitter percent, Shimmer Percent, and noise-to-harmonic ratio (NHR).
Change in Acoustic Voice Characteristics | change from 4th to the 8th dose of hormone treatment
  Digital recordings will be made using the Computerized Speech Lab (KayPENTAX) while performing the following tasks: sustained vowel /a:/, sponteous speech and "Pinokyo passage" reading. Voice recordings will be analyzed using the Real-Time Pitch Program and the Multidimensional Voice Program for measure F0, Mean F0, Jitter percent, Shimmer Percent, and noise-to-harmonic ratio (NHR).
Changes in the person's severity of depression | change from baseline to the 4th dose of hormone treatment
  - Beck depression inventory (BDI)
Changes in the person's severity of depression | change from baseline to the 8th dose of hormone treatment
  - Beck depression inventory (BDI)
Changes in the person's severity of depression | change from 4th to the 8th dose of hormone treatment
  - Beck depression inventory (BDI)
Changes in the person's perception of support | change from baseline to the 4th dose of hormone treatment
  - Multidimensional Scale of Perceived Social Support.
Changes in the person's perception of support | change from baseline to the 8th dose of hormone treatment
  - Multidimensional Scale of Perceived Social Support.
Changes in the person's perception of support | change from 4th to the 8th dose of hormone treatment
  - Multidimensional Scale of Perceived Social Support.
Changes in the person's anxiety level | change from baseline to the 4th dose of hormone treatment
  - State-trait anxiety Inventory
Changes in the person's anxiety level | change from baseline to the 8th dose of hormone treatment
  - State-trait anxiety Inventory
Changes in the person's anxiety level | change from 4th to the 8th dose of hormone treatment
  - State-trait anxiety Inventory
Changes in the person's gender perception and gender transition process | change from baseline to the 4th dose of hormone treatment
  - Transition questionnaire: The Transition Questionnaire is a self-report instrument that collects information on an individual's self-perception of status about the social and medical steps in the process of gender transition.
Changes in the person's gender perception and gender transition process | change from baseline to the 8th dose of hormone treatment
  - Transition questionnaire: The Transition Questionnaire is a self-report instrument that collects information on an individual's self-perception of status about the social and medical steps in the process of gender transition.
Changes in the person's gender perception and gender transition process | change from 4th to the 8th dose of hormone treatment
  - Transition questionnaire: The Transition Questionnaire is a self-report instrument that collects information on an individual's self-perception of status about the social and medical steps in the process of gender transition.
Changes in the person's body image perception | change from baseline to the 4th dose of hormone treatment
  -Body cathexis scale
Changes in the person's body image perception | change from baseline to the 8th dose of hormone treatment
  -Body cathexis scale
Changes in the person's body image perception | change from 4th to the 8th dose of hormone treatment
  -Body cathexis scale
Change in testosterone level | change from baseline to the 4th dose of hormone treatment
  Testosterone level measurement
Change in testosterone level | change from baseline to the 8th dose of hormone treatment
  Testosterone level measurement
Change in testosterone level | change from 4th to the 8th dose of hormone treatment
  Testosterone level measurement

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Esen AYDINLI, Assoc. Prof., Study Director — Hacettepe University, Speech and Language Therapy Departmant; Merve OGULMUS, SLP., Study Chair — Hacettepe University, Speech and Language Therapy; Koray Baser, Assoc. Prof., Study Chair — Hacettepe Univeristy, Faculty of Medicine, Mental Health and Disease Department; Bulent Okan YILDIZ, Prof., Study Chair — Hacettepe University, Faculty of Medicine, Endocrinology department; Taner YILMAZ, Prof., Study Chair — Hacettepe University, Faculty of Medicine, Otorhinolaryngology department
Locations (1):
- Hacettepe University, Speech and Language Therapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No